CLINICAL TRIAL: NCT05137379
Title: Evaluation of a Cohort of Patients With Ehlers-Danlos Syndrome Treated With Orthopedic Surgery (SED-eval)
Acronym: SED-eval
Status: Completed | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00808-31
Record Dates: First submitted 2021-10-27; First posted 2021-11-30 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2021-11

CONDITIONS: Ehlers-Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elher-Danlos syndrome patients treated with orthopedic surgery
  Interventions: Behavioral: A joint functional score based on the affected joint

INTERVENTIONS:
Behavioral: A joint functional score based on the affected joint — A joint function score according to the affected joint in patients with Ehlers-Danlos syndrome treated by surgery,: Shoulder (SSV; QuickDash), Knee (Lysholm tenger), Ankle (EFAS), Elbow and wrist (QuickDash) )

SUMMARY:
The aim of this study is to assess the joint involvement (shoulder - ankle - knee - elbow - wrist) in patients with Ehlers-Danlos Syndrome and treated by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years-old suffering from Ehlers-Danlos Syndrome and belonging to the EDS cohort of Raymond Poincaré Hospital in Garches
* Patient with joint involvement of the shoulder treated by surgery
* Patient with ankle joint damage treated by surgery
* Patient with joint damage to the knee treated by surgery
* Patient with elbow joint damage treated by surgery
* Patient with joint involvement of the wrist treated by surgery
* Patient affiliated or beneficiary of a social security scheme
* Patient who has been informed of the research and does not object to the use of his data.

Exclusion Criteria:

* Patient objecting to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years-old, suffering from Ehler-Danlos syndrome treated with surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Joint function score according to the affected joint | 1 day
  A joint function score according to the affected joint in patients with Ehlers-Danlos syndrome treated by surgery,:
  * Shoulder (SSV; QuickDash),
Joint function score according to the affected joint | 1 day
  A joint function score according to the affected joint in patients with Ehlers-Danlos syndrome treated by surgery,:
  * Knee (Lysholm tenger),
Joint function score according to the affected joint | 1 day
  A joint function score according to the affected joint in patients with Ehlers-Danlos syndrome treated by surgery,:
  * Ankle (EFAS),
Joint function score according to the affected joint | 1 day
  A joint function score according to the affected joint in patients with Ehlers-Danlos syndrome treated by surgery,:
  -Elbow and wrist (QuickDash) )

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Maussins-Nollet, Paris
  - Hôpital Raymond Poincaré, Garches, Île-de-France Region